CLINICAL TRIAL: NCT04698486
Title: Investigation of Hepatic and Cardiac Fatty Acid Metabolism in Patients With Type 2 Diabetes Mellitus With and Without Non-alcoholic Fatty Liver Disease
Brief Title: Hepatic and Cardiac Metabolic Flexibility in Subjects With T2DM With and Without NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Diabetes Academy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 74772
Record Dates: First submitted 2020-12-15; First posted 2021-01-07 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2020-12

CONDITIONS: NAFLD - Non-Alcoholic Fatty Liver Disease; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 Diabetes with NAFLD (Active Comparator): Patients with Type 2 Diabetes with NAFLD
  MR spectroscopy verified no steatosis
  Interventions: Other: Hyperinsulinemic euglycaemic clamp
- Type 2 Diabetes without NAFLD (Active Comparator): Patients with Type 2 Diabetes without NAFLD
  MR spectroscopy verified steatosis
  Interventions: Other: Hyperinsulinemic euglycaemic clamp

INTERVENTIONS:
Other: Hyperinsulinemic euglycaemic clamp — Infusion of constant intravenous insulin to achieve hyperinsulinemia and concomitant infusion of glucose to maintain euglycemia (plasma glucose at 5 mM).
  Infusion of palmitate and VLDL-triglyceride tracer. PET/CT scans of heart and liver, both in basal period and during intervention.

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) covers a spectrum from simple reversible hepatic steatosis to inflammation and fibrosis termed steatohepatitis (NASH) and cirrhosis. Accumulating evidence indicates that NAFLD is associated with development of heart failure, abnormal ventricular glucose and fatty acid (FA) utilisation and cardiac steatosis. The mechanisms behind why some subjects progress from NAFLD to NASH and the link between cardiac involvement and NAFLD are poorly understood, but must include altered cardiac and intrahepatic lipid handling. Investigators plan comprehensive kinetic studies of heart and liver FA uptake and oxidation, ventricular function and substrate utilisation, and hepatic triglyceride (TG) secretion in order to assess mechanisms governing cardiac and hepatic lipid and glucose trafficking in subjects with type 2 diabetes with and without NAFLD and NASH and the relationship with heart function. In addition, the investigators will assess skeletal muscle and adipose tissue enzyme activities, gene expression and protein concentrations in type 2 diabetic subjects to define mechanisms involved in the cross-talk between heart, liver, muscle and adipose tissues. Investigators will address these questions using tracer techniques (11Cpalmitate PET tracers and triglyceride (TG) tracers) to study cardiac and liver substrate trafficking, as well as MR spectroscopy, echocardiography, muscle and fat biopsies in combination with state-of-the art muscle and adipose tissue enzyme kinetics, gene- and protein expression. The overarching goals are to define abnormalities and differences between NAFLD and NASH in hepatic lipid (FA and TG) metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 2 Diabetes with and without NAFLD (steatosis FF% > 5,6% on MR spectroscopy for NAFLD and NASH groups)

Exclusion Criteria:

* Active smoking
* Comorbidity other than hypertension and hyperlipidemia
* Fixed medical drug consumption (including insulin) except statins and anti-diabetic medications. However, statins and weekly based GLP-1 agonist must be paused 1 week before the examination date and other antidiabetic medication 3 days before the study date.
* Patients with cancer or former cancer patients
* Blood donation within the last 3 months prior to the study
* Participation in experiments involving radioactive isotopes within the last 3 months
* Alcohol abuse (over 21 items per week for men and over 14 for women)
* Pregnancy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Fatty acid uptake in Heart (mg/kg/min) | 1 day
  Infusion of [11-C] palmitate and measured by PET/CT scan.
Fatty acid oxidation in Heart (µmol/min) | 1 day
  Infusion of [11-C] palmitate and measured by PET/CT scan.

SECONDARY OUTCOMES:
VLDL-triglyceride secretion (µmol/min) | 1 day
  Ex vivo labeled VLDL [14C]-triolein tracer technique.
VLDL-triglyceride oxidation (µmol/min) | 1 day
  Oxidation is measured by specific activity in exhaled air.
Fatty acid uptake in liver (mg/kg/min) | 1 day
  Infusion of [11-C] palmitate and measured by PET/CT scan.
Fatty acid oxidation in liver (µmol/min) | 1 day
  Infusion of [11-C] palmitate and measured by PET/CT scan.
VLDL-triglyceride uptake in muscle (percent) | 1 day
  Measurement of fatty acid concentration and specific activity in muscle biopsies
VLDL-triglyceride uptake in adipose tissue (percent) | 1 day
  Measurement of fatty acid concentration and specific activity in adipose tissue biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus N, Denmark